CLINICAL TRIAL: NCT01615185
Title: A Randomized, Double-blind, Comparison of the Efficacy and Safety of Amisulpride Versus Low-dose Amisulpride Plus Low-dose Sulpiride in the Treatment of Schizophrenia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Kai-Suan Psychiatric Hospital (Other Government)
Responsible Party: Principal Investigator, Ching-Hua Lin, MD, PhD, Chief of Adult Psychiatry, Kaohsiung Kai-Suan Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KSPH-2008-13; KSPH-2008-13
Record Dates: First submitted 2012-06-03; First posted 2012-06-08 (Estimated); Last update posted 2016-03-01 (Estimated); Status verified 2016-02

CONDITIONS: Schizophrenia
Keywords: schizophrenia; amisulpride; sulpiride; antipsychotic combination
MeSH Terms: conditions — Schizophrenia | interventions — Amisulpride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sulpiride plus amisulpride (Experimental): sulpiride 800mg/d + amisulpride 400mg/d
  Interventions: Drug: full-dose amisulpride
- full-dose amisulpride (Active Comparator): amisulpride 800mg/d
  Interventions: Drug: full-dose amisulpride

INTERVENTIONS:
Drug: full-dose amisulpride — amisulpride 800mg/d
  Other Names: Solian

SUMMARY:
Background: Surveys have shown that antipsychotic drug combinations are frequently prescribed. Amisulpride, an atypical antipsychotic agent, has low incidence of extrapyramidal symptom (EPS) but with high cost compared to sulpiride. The objective of the study is to compare the efficacy and safety of the 800-mg/d amisulpride and 400-mg/d amisulpride plus 800-mg sulpiride in the treatment of acute psychotic exacerbations of schizophrenia.

Method: In this 6-week, double-blind, fixed-dose study, patients with schizophrenia are randomly assigned to amisulpride (800 mg/d) or amisulpride (400 mg/d) plus sulpiride (800 mg/d).The hypothesis is that the two treatment groups have the similar efficacy and safety, but different cost.

DETAILED DESCRIPTION:
Background: Antipsychotic monotherapy is recognized as the treatment of choice for patients with schizophrenia. Surveys have shown that antipsychotic drug combinations are frequently prescribed, yet few clinical studies have examined this practice. Amisulpride, an atypical antipsychotic agent, has low incidence of extrapyramidal symptom (EPS) but with high cost compared to sulpiride. It has been reported that mean doses of low-potency typical antipsychotics less than 600 mg/day of chlorpromazine equivalent dose has no higher risk of EPS than atypical antipsychotics. The objective of the study is to compare the efficacy and safety of the 800-mg/d amisulpride and 400-mg/d amisulpride plus 800-mg sulpiride in the treatment of acute psychotic exacerbations of schizophrenia.

Method: In this 6-week, double-blind, fixed-dose study, patients with schizophrenia (DSM-IV diagnosis) are randomly assigned to amisulpride (800 mg/d) or amisulpride (400 mg/d) plus sulpiride (800 mg/d). The hypothesis is that the two treatment groups have the similar efficacy and safety, but different cost. The efficacy assessment was the change from baseline in the score on the Clinical Global Impression-Severity (CGI-S), Positive and Negative Syndrome Scale (PANSS) and subscales (positive scale, negative scale, general psychopathology scale), Calgary Depression Scale for Schizophrenia (CDSS), and Global Assessment of Functioning (GAF). Safety assessments include the change from baseline on Simpson-Angus Rating Scale (SAS), Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Scale (BAS), and UKU Side-effects Rating Scale (UKU), and the change from baseline in prolactin levels, body weight, vital sign, blood pressure, AC glucose level, and lipid profiles(cholesterol, high density lipid protein [HDL], low density lipid protein [LDL], and triglyceride [TG]).

ELIGIBILITY:
Inclusion Criteria:

* schizophrenia
* CGI >=4
* washout of antipsychotics at least 3-5 days
* written informed consents

Exclusion Criteria:

* History of serious adverse events to sulpiride or amisulpride
* History of neuroleptic malignant syndrome or tardive dyskinesia to antipsychotics
* treatment-resistant schizophrenia
* long-acting antipsychotics in the past 3 months
* comorbid with substance abuse/dependence
* female subjects with pregnancy
* severe physical illness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Actual)
Dates: Start 2008-01; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
change from baseline in Positive and Negative Syndrome Scale (PANSS) total scores | The PANSS was rated at baseline, and again at weeks 1, 2, 3, 4, and 6 (or on early termination).

SECONDARY OUTCOMES:
changes from baseline in the scores on several psychopathology scales for efficacy | The CGI-S, PANSS, CDSS, and GAF were rated at baseline, and again at weeks 1, 2, 3, 4, and 6 (or on early termination).
  psychopathology scales for efficacy include: Clinical Global Impression-Severity (CGI-S), PANSS positive scale, PANSS negative scale, PANSS general psychopathology scale, Calgary Depression Scale for Schizophrenia (CDSS), and Global Assessment of Functioning (GAF)
Assessments of safety for extrapyramidal symptoms (EPS) | AIMS, BAS, and SAS were administered at baseline and at weeks 1, 2, 3, 4, and 6 (or on early termination)
  The severity of EPS was assessed by the following neurological scales: the Abnormal Involuntary Movement Scale (AIMS), Barnes Akathisia Scale (BAS), and the Simpson-Angus Rating Scale (SAS)
Assessments of safety for general adverse events | UKU was administered at baseline and at weeks 1, 2, 3, 4, and 6 (or on early termination)
  General adverse events were evaluated by a standardized the UKU Side Effect Rating Scale. A score of 1, 2 or 3 on any UKU item that first occurred or worsened during treatment indicated adverse events "cases".
Other safety of clinical trial | Body weight, BMI, pulse rate, and blood pressure were checked at baseline and at weeks 1, 2, 3, 4, and 6 (or on early termination). ECG and laboratory tests were assessed at baseline and week 6.
  Body weights, body mass index (BMI), pulse rate, blood pressure (systolic and diastolic), 12-lead electrocardiogram (ECG) for QTc intervals (Bazett's correction of QT interval), and laboratory tests were performed to determine safety. Laboratory tests included fasting glucose, liver function (alanine aminotransferase [ALT] and aspartate aminotransferase [AST]), renal function (blood urea nitrogen [BUN], creatinine), lipid profiles (triglycerides, cholesterol, high density lipoprotein [HDL], and low density lipoprotein [LDL]), and prolactin level.
Assessments of quality of life | Medical Outcomes Study Short-Form 36 was assessed at baseline and week 6
  The SF-36, with two primary-factor analytic components: the physical component summary and the mental component summary, was used to measure quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hua Lin, MD, PhD, Principal Investigator — Kai-Suan Psychiatric Hospital
Locations (1):
- Kai-Suan Psychiatric Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Result] Leucht S, Wahlbeck K, Hamann J, Kissling W. New generation antipsychotics versus low-potency conventional antipsychotics: a systematic review and meta-analysis. Lancet. 2003 May 10;361(9369):1581-9. doi: 10.1016/S0140-6736(03)13306-5. PMID 12747876
- [Result] Kapur S, Seeman P. Does fast dissociation from the dopamine d(2) receptor explain the action of atypical antipsychotics?: A new hypothesis. Am J Psychiatry. 2001 Mar;158(3):360-9. doi: 10.1176/appi.ajp.158.3.360. PMID 11229973
- [Result] McKeage K, Plosker GL. Amisulpride: a review of its use in the management of schizophrenia. CNS Drugs. 2004;18(13):933-56. doi: 10.2165/00023210-200418130-00007. PMID 15521794
- [Result] Chakos MH, Glick ID, Miller AL, Hamner MB, Miller DD, Patel JK, Tapp A, Keefe RS, Rosenheck RA. Baseline use of concomitant psychotropic medications to treat schizophrenia in the CATIE trial. Psychiatr Serv. 2006 Aug;57(8):1094-101. doi: 10.1176/ps.2006.57.8.1094. PMID 16870959
- [Derived] Lin CH, Wang FC, Lin SC, Huang YH, Chen CC, Lane HY. Antipsychotic combination using low-dose antipsychotics is as efficacious and safe as, but cheaper, than optimal-dose monotherapy in the treatment of schizophrenia: a randomized, double-blind study. Int Clin Psychopharmacol. 2013 Sep;28(5):267-74. doi: 10.1097/YIC.0b013e3283633a83. PMID 23778382